CLINICAL TRIAL: NCT05199870
Title: Post-Market Clinical Follow-Up Study to Provide Safety, Performance and Clinical Benefits Data of the RingLoc Bipolar Acetabular Cup or Endo II Heads (Implants and Instrumentation) in Hip Hemiarthroplasty - A Retrospective Enrollment/Prospective Follow-Up Consecutive Series Study
Brief Title: MDR - PMCF Study for RingLoc Bipolar Acetabular Cup and Endo II Femoral Heads
Status: Not yet recruiting | Type: Observational
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: MDRG2017-89MS-43H
Record Dates: First submitted 2022-01-05; First posted 2022-01-20 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Hip Arthritis; Hip Disease; Hip Fractures; Hip Injuries; Hip Pain Chronic
MeSH Terms: conditions — Hip Fractures; Hip Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- RingLoc Bipolar Acetabular Cup: Patients that have been implanted with the RingLoc Bipolar acetabular cup to repair hip malfunction/disease/injury.
  Interventions: Device: RingLoc Bipolar Acetabular Cup
- Endo II Femoral Heads: Subjects who were implanted with the Endo II Femoral head during hemiarthroplasty
  Interventions: Device: Endo II Femoral Head

INTERVENTIONS:
Device: RingLoc Bipolar Acetabular Cup — Patients that have been implanted with a RingLoc Bipolar acetabular cup.
  Groups: RingLoc Bipolar Acetabular Cup
Device: Endo II Femoral Head — Subjects that have been implanted with an Endo II Femoral Head
  Groups: Endo II Femoral Heads

SUMMARY:
The objective of this retrospective enrollment/prospective follow-up consecutive series PMCF study is to collect data confirming safety, performance, and clinical benefits of the RingLoc Bipolar Acetabular Cup and the Endo II Femoral Head when used for hip hemiarthroplasty (implants and instrumentation).

DETAILED DESCRIPTION:
The objective of this retrospective enrollment/prospective follow-up consecutive series PMCF study is to collect data confirming safety, performance, and clinical benefits of the RingLoc Bipolar Acetabular Cup and the Endo II Femoral Head when used for hip hemiarthroplasty (implants and instrumentation).

The primary objective of this study is the assessment of safety by analyzing implant survivorship at the longest follow-up timepoint available, greater than or equal to eight years post-implantation. This will be established by recording the incidence and frequency of revisions, complications, and adverse events. Relationship of the events to implant, instrumentation and/or procedure should be specified.

The secondary objective is the assessment of performance and clinical benefits by recording patient-reported clinical outcomes measures (PROMs).

ELIGIBILITY:
Inclusion Criteria:

* Patient must be 18 years of age or older and skeletally mature
* Patient must have undergone hip hemiarthroplasty surgery with the RingLoc Bipolar Acetabular Cup or Endo II Femoral Head for a cleared indication, greater than or equal to eight years previous to the date of study consent. Cleared indications for the RingLoc Bipolar and Endo II Heads include the following:

  * Noninflammatory degenerative joint disease including osteoarthritis and avascular necrosis
  * Rheumatoid arthritis
  * Correction of functional deformity
  * Treatment of non-union, femoral neck fracture, and trochanteric fractures of the proximal femur with head involvement, unmanageable using other techniques.

Exclusion Criteria:

* Any medical diagnosis present at the time of surgery that, at the Investigator's discretion, could compromise the implant's survivability
* Off-label use or not according to the approved instructions for use (IFU) of study devices
* Revision procedures where other treatment or devices have failed
* Uncooperative patient or patient with neurologic disorders who is incapable of following directions
* Patient has a psychiatric illness or

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A consecutive series of patients implanted with the RingLoc Bipolar acetabular cup or the Endo II Femoral Head.
Sampling Method: Non-Probability Sample
Enrollment: 116 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2030-09-03 (Estimated); Study Completion 2030-09-03 (Estimated)

PRIMARY OUTCOMES:
Device safety assessed through the frequency and incidence of revisions, complications, and Adverse Events. | Greater than or equal to 8 years.
  The primary objective of this study is the assessment of safety by analyzing implant survivorship. This will be established by recording the incidence and frequency of revisions, complications, and Adverse Events. Relation of the events to either implant or instrumentation will be specified.

SECONDARY OUTCOMES:
Device Performance and Benefits evaluated through the Oxford Hip Score and Patient Assessment. | Greater than or equal to 8 years.
  The OHS is a patient-completed, 12-question evaluation. Each item is scored from 1 to 5, with 1 representing best outcome/least symptoms and 5 representing worst outcome/most symptoms. The Patient Assessment is patient completed and a 4-question evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Lynsey Boyle, Study Director — Zimmer Biomet
Locations (1):
- Inova Fairfax Hospital, Falls Church, Virginia, United States

IPD SHARING:
Plan to Share IPD: No